CLINICAL TRIAL: NCT03283709
Title: Removable Partial Denture Abutments Restored With Monolithic Zirconia Crowns: A Randomized Controlled Trial
Brief Title: Removable Partial Denture Abutments Restored With Monolithic Zirconia Crowns
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated because PI left the institution.
Sponsor: Hiroko Nagaoka (Other)
Responsible Party: Sponsor-Investigator, Hiroko Nagaoka, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0511-F1V
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Crowns; Denture

STUDY DESIGN:
Intervention Model Description: A prospective, randomized controlled trial comparing treatment outcomes for partial edentulism using two restorative materials. A convenience sample of study participants will be randomly assigned to either a treatment group or a control group.
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Full-contour monolithic Zirconia crowns (Experimental): If participants assigned to this arm are in need of surveyed crowns on RPD abutment teeth they will be fabricated from multi-layered monolithic zirconia
  Interventions: Device: Full-contour monolithic zirconia abutment crowns
- Conventional abutment crowns (Other): If participants assigned to this arm are in need of surveyed crowns on RPD abutment teeth they will be fabricated from type III gold or high-noble metal veneered with feldspathic porcelain
  Interventions: Device: Conventional abutment crowns

INTERVENTIONS:
Device: Full-contour monolithic zirconia abutment crowns — Subjects with RPD abutment teeth that require surveyed crowns will have them fabricated from monolithic multi-layered zirconia
  Arms: Full-contour monolithic Zirconia crowns
Device: Conventional abutment crowns — Subjects with RPD abutment teeth that require surveyed crowns will have them fabricated from noble or high noble metals, veneered with feldspathic porcelain
  Arms: Conventional abutment crowns

SUMMARY:
The purpose of this study is to investigate the use of an all-ceramic dental crown material to restore the abutment teeth of partially-edentulous patients who need removable partial dentures (RPD). The outcomes of the treatment group (all-ceramic crowns) will be compared to a similarly-treated control group whose RPD abutment teeth are restored using conventional metal and metal-ceramic crowns. Primary outcomes of interest include crown survival, abutment tooth survival and RPD survival.The null hypothesis is that at the conclusion of the study there will be no differences in outcomes between the two groups.

All dental treatment, including dental hygiene and periodontal care, fillings, crowns and RPD fabrication will be provided by predoctoral dental students in the University of Kentucky College of Dentistry student clinics. Students treating the subjects will be supervised by licensed, technique-calibrated faculty specialists. Following the completion of dental treatment, enrolled subjects will be clinically re-evaluated by investigators at 6 months, and at annual intervals thereafter for 5 years following RPD delivery.

DETAILED DESCRIPTION:
This study will investigate the use of highly esthetic, second and third generation multi-layer zirconia crown materials to restore removable partial denture abutment teeth. All performed treatment will be the standard of care and to the usual and customary standards used in United states dental clinics for crown and RPD procedures. Treatment subjects will have RPD abutment teeth restored with either Noritake Katana STML (anterior teeth) or HTML (premolars and molars) zirconia crowns, and periodically evaluated for 60 months following RPD delivery. Outcomes will be compared to a similarly treated control group restored with metal, metal-ceramic, or a combination of metal and metal-ceramic crowns.

Following informed consent, subjects will be randomly assigned using an internet program (https://www.randomizer.org/) to either a treatment (zirconia abutment tooth crown) or control (metal or metal-ceramic abutment tooth crown) group. Using information from the oral examination, articulated diagnostic casts will be evaluated , the RPD design confirmed, and the need for a crown on one or more abutment teeth verified. Enrolled subjects will be given oral hygiene instruction at the beginning of the study. They will also be instructed to brush their teeth twice daily using an OTC fluoride dentifrice of their choice. They will also be asked to use a 0.05% NaF oral rinse for 1 minute daily.

Abutment teeth must be in function with the opposing arch and vital at the beginning of the study. Vitality will be be determined using a synthesis of history, percussion, palpation and pulp testing. Pulp tests will be conducted using cold and an EPT, and the facial, lingual and occlusal (incisal) surfaces of all abutment teeth will be tested for responsiveness. If abutment tooth vitality is confirmed, teeth requiring surveyed crowns will be prepared and restored using standardized clinical and laboratory guidelines.

Abutment teeth restored with metal and zirconia crowns will be prepared and restored using the following clinical and laboratory guidelines. The margin will be a circumferential chamfer prepared to a depth of 0.5 mm with a rounded internal line angle and a 90° cavosurface exit angle. Margin height will be at or slightly coronal to the free gingival margin where possible. Axial surfaces will be prepared with a total occlusal convergence of >6° but not to exceed 20°. Incisal and facial surfaces will be reduced 0.7-1.0 mm. Functional surfaces will be reduced to 1.0 mm of opposing tooth clearance with the exception of under rest seats, where opposing tooth clearance will be 2.0 mm. At completion, the prepared tooth should have a height to base ratio of 0.4. If inadequate retention and resistance form is identified following preparation of axial walls, supplementary grooves will be added, the number and location of which are at the discretion of the investigator. Final impressions will be made using PVS in a custom tray (Extrude) and poured in type V dental stone (Jadestone). Following fabrication, the working cast will be articulated, tripoded, and the die(s) sectioned, trimmed and scanned (3Shape D2000 laboratory scanner or equivalent). The crown(s) will be waxed to full contour. Rest seats, undercuts and guide planes will then be developed in wax. Once the waxup has been surveyed and finalized, it will be secured to the scanning platform and a new scan performed with the waxup in place. The data file with the die scan will be merged with the file that contains the waxup. The merged file will then be transmitted to a designated production facility where the zirconia crown(s) will be milled. Canines will be milled using Noritake Katana STML zirconia and premolars and molars will be milled using Noritake Katana HTML zirconia. Once the crown(s) are returned and the margins, contacts, occlusion and contours clinically verified, they will be luted using a self-adhesive resin-based cement (RelyX Unicem 2).

Porcelain-fused-to-metal (PFM) crowns will be prepared and restored using a standard protocol utilizing the following guidelines. Posterior crowns will have metal occlusal surfaces with the porcelain-metal junction on the occlusal surface at half the distance between the central groove and the buccal cusp tip. Mesial, distal and lingual surfaces will be in metal, and the crown will have a disappearing metal margin on the facial surface. The facial preparation from mesiofacial to distofacial line angles will be a heavy chamfer or modified shoulder 1.0-1.2 mm in depth with a rounded internal line angle and a 90° cavosurface exit angle. Mesial, distal and lingual chamfer margins will be prepared to a horizontal depth of 0.5 mm. Facial margin height will be at or slightly apical to the free gingival margin. Mesial, distal and lingual margin height will be at or slightly coronal to the free gingival margin if possible. Functional surfaces will be prepared with opposing tooth clearance of 1.5 mm with the exception of under rest seats where opposing tooth clearance will be 2.0 mm. Nonfunctional cusp reduction will be 1.0 mm. Final impressions will be made using PVS (Extrude) in a custom tray and poured in type V dental stone (Jadestone). Following working cast fabrication it will be articulated, tripoded, and the die(s) prepared for conventional laboratory crown fabrication. Conventional (all-metal and PFM) surveyed crowns will be fabricated using noble and high-noble casting alloys and PFM crowns will use feldspathic porcelain as a veneering ceramic. Once the crown(s) are returned and the margins, contacts, occlusion and contours clinically verified, they will be luted using a self-adhesive resin-based cement (RelyX Unicem 2).

Qualifying RPD designs may be Kennedy class I-IV with up to two modification spaces, and will be designed using a standardized protocol. Maxillary major connectors may consist of a complete palatal plate, modified palatal plate, anterior-posterior palatal strap or palatal strap. Mandibular major connectors will consist of either a lingual plate or a lingual bar. Frameworks will be fabricated from nickel-chrome alloy (Ticonium), the denture bases acrylic resin (Lucitone 199), and artificial teeth will be DENTSPLY Trubyte IPN Portrait. To meet the definition of an RPD abutment tooth it must host a direct retainer consisting of an occlusal or cingulum rest, a proximal plate and a retentive clasp. Reciprocation must be provided in the form of a plate, reciprocating clasp or minor connector and rest. The plan for occlusion will be based upon the number and distribution of remaining natural teeth. If an arch opposing the RPD is edentulous and restored by a removable complete denture, then natural and artificial teeth will be arranged in bilateral balance. If anterior guidance is present on natural teeth in both arches it will be preserved so that artificial RPD teeth contact opposing teeth in maximum intercuspation only.

Clinical assessments, procedures and annual examinations will be performed in the University of Kentucky College of Dentistry second, third, and fourth floor student clinics. Clinical procedures will be performed by third and fourth year dental students, and clinical supervision for these procedures will be provided by licensed, calibrated investigators.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous and treatment planned for an RPD
* Requires at least 1 surveyed crown on an abutment tooth
* Abutment teeth and RPD in function with opposing arch
* Abutment teeth vital at time of study enrollment
* English literacy, cognitively capable of understanding study and consent documents
* Cognitively and functionally capable of performing prosthesis and oral self-care

Exclusion Criteria:

* Any chronic or degenerative condition which impairs consent capability
* Any cognitive or motor condition which impairs ability to follow instructions or perform oral self-care
* Healthy enough to tolerate planned dental procedures without premedication
* Chronic infectious disease
* COPD
* Renal insufficiency
* Autoimmune or chronic inflammatory disorders
* Unstable asthma or diabetes
* Unstable hypertension

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaughan Hoefler, DDS, MBA, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky College of Dentistry, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Douglass CW, Watson AJ. Future needs for fixed and removable partial dentures in the United States. J Prosthet Dent. 2002 Jan;87(1):9-14. doi: 10.1067/mpr.2002.121204. PMID 11807477
- [Background] Campbell SD, Cooper L, Craddock H, Hyde TP, Nattress B, Pavitt SH, Seymour DW. Removable partial dentures: The clinical need for innovation. J Prosthet Dent. 2017 Sep;118(3):273-280. doi: 10.1016/j.prosdent.2017.01.008. Epub 2017 Mar 23. PMID 28343666
- [Background] Abt E, Carr AB, Worthington HV. Interventions for replacing missing teeth: partially absent dentition. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD003814. doi: 10.1002/14651858.CD003814.pub2. PMID 22336794
- [Background] Benso B, Kovalik AC, Jorge JH, Campanha NH. Failures in the rehabilitation treatment with removable partial dentures. Acta Odontol Scand. 2013 Nov;71(6):1351-5. doi: 10.3109/00016357.2013.777780. Epub 2013 Jul 9. PMID 23834529
- [Background] Ettinger RL, Goettsche ZS, Qian F. The Extent and Scope of Prosthodontic Practice in Iowa. J Prosthodont. 2019 Feb;28(2):113-121. doi: 10.1111/jopr.12588. Epub 2017 Mar 8. PMID 28273692
- [Background] Rehmann P, Orbach K, Ferger P, Wostmann B. Treatment outcomes with removable partial dentures: a retrospective analysis. Int J Prosthodont. 2013 Mar-Apr;26(2):147-50. doi: 10.11607/ijp.2959. PMID 23476909
- [Background] De Kok IJ, Cooper LF, Guckes AD, McGraw K, Wright RF, Barrero CJ, Bak SY, Stoner LO. Factors Influencing Removable Partial Denture Patient-Reported Outcomes of Quality of Life and Satisfaction: A Systematic Review. J Prosthodont. 2017 Jan;26(1):5-18. doi: 10.1111/jopr.12526. Epub 2016 Sep 6. PMID 27598416
- [Background] Murai S, Matsuda K, Ikebe K, Enoki K, Hatta K, Fujiwara K, Maeda Y. A field survey of the partially edentate elderly: Investigation of factors related to the usage rate of removable partial dentures. J Oral Rehabil. 2015 Nov;42(11):828-32. doi: 10.1111/joor.12318. Epub 2015 Jun 7. PMID 26059645
- [Background] Koyama S, Sasaki K, Yokoyama M, Sasaki T, Hanawa S. Evaluation of factors affecting the continuing use and patient satisfaction with Removable Partial Dentures over 5 years. J Prosthodont Res. 2010 Apr;54(2):97-101. doi: 10.1016/j.jpor.2009.11.007. Epub 2010 Jan 18. PMID 20083450
- [Background] Raigrodski AJ. Contemporary materials and technologies for all-ceramic fixed partial dentures: a review of the literature. J Prosthet Dent. 2004 Dec;92(6):557-62. doi: 10.1016/j.prosdent.2004.09.015. PMID 15583562
- [Background] Donovan TE. Factors essential for successful all-ceramic restorations. J Am Dent Assoc. 2008 Sep;139 Suppl:14S-18S. doi: 10.14219/jada.archive.2008.0360. PMID 18768904
- [Background] Kelly JR. Dental ceramics: what is this stuff anyway? J Am Dent Assoc. 2008 Sep;139 Suppl:4S-7S. doi: 10.14219/jada.archive.2008.0359. No abstract available. PMID 18768902
- [Background] Spear F, Holloway J. Which all-ceramic system is optimal for anterior esthetics? J Am Dent Assoc. 2008 Sep;139 Suppl:19S-24S. doi: 10.14219/jada.archive.2008.0358. PMID 18768905
- [Background] Sailer I, Makarov NA, Thoma DS, Zwahlen M, Pjetursson BE. All-ceramic or metal-ceramic tooth-supported fixed dental prostheses (FDPs)? A systematic review of the survival and complication rates. Part I: Single crowns (SCs). Dent Mater. 2015 Jun;31(6):603-23. doi: 10.1016/j.dental.2015.02.011. Epub 2015 Apr 2. PMID 25842099
- [Background] Larsson C, Wennerberg A. The clinical success of zirconia-based crowns: a systematic review. Int J Prosthodont. 2014 Jan-Feb;27(1):33-43. doi: 10.11607/ijp.3647. PMID 24392475
- [Background] Le M, Papia E, Larsson C. The clinical success of tooth- and implant-supported zirconia-based fixed dental prostheses. A systematic review. J Oral Rehabil. 2015 Jun;42(6):467-80. doi: 10.1111/joor.12272. Epub 2015 Jan 10. PMID 25580846
- [Background] Ozkurt Z, Kazazoglu E. Clinical success of zirconia in dental applications. J Prosthodont. 2010 Jan;19(1):64-8. doi: 10.1111/j.1532-849X.2009.00513.x. Epub 2009 Sep 14. PMID 19754642
- [Background] Ozer F, Mante FK, Chiche G, Saleh N, Takeichi T, Blatz MB. A retrospective survey on long-term survival of posterior zirconia and porcelain-fused-to-metal crowns in private practice. Quintessence Int. 2014 Jan;45(1):31-8. doi: 10.3290/j.qi.a30768. PMID 24392493
- [Background] Burns DR, Unger JW. The construction of crowns for removable partial denture abutment teeth. Quintessence Int. 1994 Jul;25(7):471-5. PMID 7991768
- [Background] Kancyper S, Sierraalta M, Razzoog ME. All-ceramic surveyed crowns for removable partial denture abutments. J Prosthet Dent. 2000 Oct;84(4):400-2. doi: 10.1067/mpr.2000.110253. PMID 11044845
- [Background] Carracho JF, Razzoog ME. Removable partial denture abutments restored with all-ceramic surveyed crowns. Quintessence Int. 2006 Apr;37(4):283-8. PMID 16594359
- [Background] Yoon TH, Chang WG. The fabrication of a CAD/CAM ceramic crown to fit an existing partial removable dental prosthesis: a clinical report. J Prosthet Dent. 2012 Sep;108(3):143-6. doi: 10.1016/S0022-3913(12)60137-1. PMID 22944309
- [Background] Pihlaja J, Napankangas R, Kuoppala R, Raustia A. Veneered zirconia crowns as abutment teeth for partial removable dental prostheses: a clinical 4-year retrospective study. J Prosthet Dent. 2015 Nov;114(5):633-6. doi: 10.1016/j.prosdent.2015.05.008. Epub 2015 Sep 4. PMID 26346419
- [Background] Denry I, Kelly JR. Emerging ceramic-based materials for dentistry. J Dent Res. 2014 Dec;93(12):1235-42. doi: 10.1177/0022034514553627. Epub 2014 Oct 1. PMID 25274751
- [Background] Johansson C, Kmet G, Rivera J, Larsson C, Vult Von Steyern P. Fracture strength of monolithic all-ceramic crowns made of high translucent yttrium oxide-stabilized zirconium dioxide compared to porcelain-veneered crowns and lithium disilicate crowns. Acta Odontol Scand. 2014 Feb;72(2):145-53. doi: 10.3109/00016357.2013.822098. Epub 2013 Jul 18. PMID 23865549
- [Background] Stober T, Bermejo JL, Rammelsberg P, Schmitter M. Enamel wear caused by monolithic zirconia crowns after 6 months of clinical use. J Oral Rehabil. 2014 Apr;41(4):314-22. doi: 10.1111/joor.12139. Epub 2014 Jan 22. PMID 24447258
- [Background] Flinn BD, Raigrodski AJ, Mancl LA, Toivola R, Kuykendall T. Influence of aging on flexural strength of translucent zirconia for monolithic restorations. J Prosthet Dent. 2017 Feb;117(2):303-309. doi: 10.1016/j.prosdent.2016.06.010. Epub 2016 Sep 22. PMID 27666494
- [Background] Sulaiman TA, Abdulmajeed AA, Donovan TE, Ritter AV, Vallittu PK, Narhi TO, Lassila LV. Optical properties and light irradiance of monolithic zirconia at variable thicknesses. Dent Mater. 2015 Oct;31(10):1180-7. doi: 10.1016/j.dental.2015.06.016. Epub 2015 Jul 18. PMID 26198027
- [Background] Harada K, Raigrodski AJ, Chung KH, Flinn BD, Dogan S, Mancl LA. A comparative evaluation of the translucency of zirconias and lithium disilicate for monolithic restorations. J Prosthet Dent. 2016 Aug;116(2):257-63. doi: 10.1016/j.prosdent.2015.11.019. Epub 2016 Mar 17. PMID 26994676
- [Background] Sulaiman TA, Abdulmajeed AA, Donovan TE, Cooper LF, Walter R. Fracture rate of monolithic zirconia restorations up to 5 years: A dental laboratory survey. J Prosthet Dent. 2016 Sep;116(3):436-9. doi: 10.1016/j.prosdent.2016.01.033. Epub 2016 May 11. PMID 27178771
- [Background] Belli R, Petschelt A, Hofner B, Hajto J, Scherrer SS, Lohbauer U. Fracture Rates and Lifetime Estimations of CAD/CAM All-ceramic Restorations. J Dent Res. 2016 Jan;95(1):67-73. doi: 10.1177/0022034515608187. Epub 2015 Oct 1. PMID 26428908
- [Background] Batson ER, Cooper LF, Duqum I, Mendonca G. Clinical outcomes of three different crown systems with CAD/CAM technology. J Prosthet Dent. 2014 Oct;112(4):770-7. doi: 10.1016/j.prosdent.2014.05.002. Epub 2014 Jun 28. PMID 24980739
- [Background] Ueda K, Guth JF, Erdelt K, Stimmelmayr M, Kappert H, Beuer F. Light transmittance by a multi-coloured zirconia material. Dent Mater J. 2015;34(3):310-4. doi: 10.4012/dmj.2014-238. Epub 2015 Apr 23. PMID 25904173
- [Background] Nordahl N, Vult von Steyern P, Larsson C. Fracture strength of ceramic monolithic crown systems of different thickness. J Oral Sci. 2015 Sep;57(3):255-61. doi: 10.2334/josnusd.57.255. PMID 26369491
- [Background] Stawarczyk B, Keul C, Eichberger M, Figge D, Edelhoff D, Lumkemann N. Three generations of zirconia: From veneered to monolithic. Part II. Quintessence Int. 2017;48(6):441-450. doi: 10.3290/j.qi.a38157. PMID 28497132
- [Background] Slade GD, Spencer AJ. Development and evaluation of the Oral Health Impact Profile. Community Dent Health. 1994 Mar;11(1):3-11. PMID 8193981
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Started | 0 | 1
Completed | 0 | 0
Not Completed | 0 | 1
Not completed — trial terminated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Trial was terminated early with only participant enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 1 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Need to Replace Crown on RPD Abutment Tooth
Description: This is a collective measure reporting need to replace an abutment tooth crown for any reason. This includes repeated adhesive failure at crown interface due to inadequate retention/resistance form in the abutment tooth preparation, catastrophic fracture of monolithic or veneering crown ceramic necessitating crown replacement, primary or secondary caries involving crowned abutment tooth necessitating crown replacement
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: RPD Abutment Tooth Loss
Description: Loss of any RPD abutment tooth for any reason whether crowned or otherwise.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: RPD Failure
Description: Any technical or biologic complication resulting in loss of service of RPD. This includes loss of RPD as well as dissatisfaction and nonacceptance
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Tooth Loss
Description: Loss of any nonabutment tooth in either arch for any reason
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Caries
Description: Dental caries involving any tooth in either arch
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Periodontal Disease
Description: Change in clinical attachment level involving any tooth in either arch compared to baseline presentation.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Periodontal Disease
Description: Increase or decrease in mobility involving any tooth in either arch compared to baseline presentation.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Periodontal Disease
Description: Onset of fremitus involving any tooth in either arch relative to baseline presentation.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Periodontal Disease
Description: Change in furcation classification involving any molar in either arch relative to baseline presentation..
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Periodontal Disease
Description: Change in overall score for bleeding index compared to baseline presentation.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Periodontal Disease
Description: Change in overall score for plaque index compared to baseline presentation.
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Abutment Tooth Vitality
Description: Loss of vitality of any abutment tooth, crowned or otherwise
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Patient Satisfaction and Quality of Life
Description: Change in patient satisfaction and quality of life, measured using the OHIP-14 questionnaire
Time Frame: 60 months
Population: The single enrolled participant did not complete the intervention; thus, no data were generated.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 month
Description: No participant completed the entire intervention due to trial termination (unrelated to adverse events). Thus, there are no adverse event or mortality data to report.
Arm/Group | Full-contour Monolithic Zirconia Crowns | Conventional Abutment Crowns
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03283709/Prot_SAP_000.pdf
  • Informed Consent Form (2016-02-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT03283709/ICF_001.pdf